CLINICAL TRIAL: NCT00116922
Title: CAnadian Normoglycemia Outcomes Evaluation Study
Brief Title: A Lifestyle and Combination Medication Therapy Diabetes Prevention Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CANOE
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Impaired Glucose Tolerance; Diabetes
Keywords: Diabetes; Prevention.; Rosiglitazone; Metformin; Lifestyle; Impaired glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — rosiglitazone-metformin combination; Rosiglitazone; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator): Avandamet [ Rosuglitazone 2 and Metformin 500]
  Interventions: Drug: Avandamet [Rosiglitazone 2mg/Metformin 500mg] BID

INTERVENTIONS:
Drug: Avandamet [Rosiglitazone 2mg/Metformin 500mg] BID — [Rosiglitazone 2mg/ Metformin 500mg] twice daily
  Other Names: Avandamet

SUMMARY:
It is now well established that the 21st century will be characterized by a global epidemic of Type 2 diabetes. The principal aim of the CANOE study is to determine whether individuals with the pre-diabetes condition impaired glucose tolerance can be prevented from progressing to diabetes with a healthy living lifestyle intervention and an insulin sensitizing medication. Individuals who have impaired glucose tolerance (IGT) determined during an oral glucose tolerance test will be eligible to participate in this study. All participants will receive a lifestyle dietary and exercise intervention program. Half of the participants will be randomly assigned to an insulin sensitizing medication (rosiglitazone/metformin) which is commonly used to treat Type 2 diabetes. The primary outcome for this study is the development of diabetes. The study is expected to last a total of five years.

DETAILED DESCRIPTION:
The CANOE Study CAnadian Normoglycemia Outcomes Evaluation Study

It is now well accepted that the 21st Century will be characterized by a global epidemic of Type 2 diabetes mellitus [Type 2DM]. To deal with this major health crisis, several strategies have been proposed. These include efforts that focus on the primary prevention of diabetes, attempts at implementing effective management of diabetes once it develops, and the institution of appropriate proven therapies for established diabetic complications. The CANOE study focuses on a primary prevention strategy. The study is designed to evaluate the effect of pharmacological therapy combined with a healthy living lifestyle intervention on Canadian individuals who are at high risk for this metabolic condition because they have IGT.

OBJECTIVES

* To determine if treatment with Avandamet, in addition to a healthy living lifestyle program, will prevent the development of Type 2 diabetes in Canadians at high risk for this metabolic disorder;
* To determine if treatment with Avandamet, in addition to a healthy living lifestyle program will improve cardiovascular risk factors associated with IGT.

STUDY DESIGN

CANOE is a moderately sized, randomized, double-blind controlled trial to determine if Avandamet will decrease the development of diabetes in individuals at high risk for this condition. A total of 200 patients will be followed for an average follow up of 4 years (range 3 - 5 years). Active treatment with Avandamet (Metformin 500 mg / Rosiglitazone 2 mg) administered as one capsule twice daily will be compared to matched placebo.

All study participants will receive a lifestyle intervention program based on the latest national evidence-based guidelines recommended by the Canadian Diabetes Association (Can J Diabetes, Vol 27 Suppl 2, 2003).

ELIGIBILITY:
Inclusion Criteria:

* Residents of Ontario
* Age 18-75
* IGT on OGTT

Exclusion Criteria:

* Current use of Metformin or Rosiglitazone
* Prior use of medication to treat diabetes except gestational diabetes
* Use of drugs known to exacerbate glucose tolerance
* History of diabetes except gestational diabetes
* Liver function studies greater the 2.5x normal
* Creatinine clearance less than 60 ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2004-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Development of diabetes based on 1 positive OGTT or 2 fasting glucose levels | Dec 2009

SECONDARY OUTCOMES:
Lipids, CBC, CRP, homocysteine, adiponectin, insulin, proinsulin, and routine biochemistry will be done annually | Dec2009

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Zinman, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Stewart Harris, MD, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - UWO Research Park, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario